CLINICAL TRIAL: NCT00155415
Title: A Prospective Single-Blinded Randomized Trial Comparing Colonoscopic Preparation at Different Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 9461700305
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-12-02 (Estimated); Status verified 2005-09

CONDITIONS: Colonoscopy; Colon Neoplasm
Keywords: Colonoscopy; Polyethylene glycol(PEG); Colon neoplasm; Colon cleansing; Timing
MeSH Terms: conditions — Colonic Neoplasms

INTERVENTIONS:
Behavioral: Different timing of taking polyethylene glycol(PEG)

SUMMARY:
Colorectal cancer (CRC) is the leading cause of cancer death not only in the Western countries but also in Taiwan. Colonoscopy is now gradually accepted as one of the powerful tool for colorectal cancer screening. Not only for survey after positive fecal test, it is also applied as primary screening modality for CRC screening.Colon cleansing before colonoscopy thus becomes critically important and inadequate preparation may lead to low diagnostic yield with missed lesions, increased risk of complication and prolonged procedure time. Though the importance of good colon preparation can not be over-emphasized, diet control before colonoscopy and ingestion of large amount of lavage solution remain a significant hurdle to overcome and investigators continue to seek for the ideal colon preparation with respect to quality and examinee satisfaction. After the introduction of polyethylene glycol electrolyte lavage solution (PEG-ELS) for bowel preparation before colon procedures, its safety was well documented and the efficacy of colon cleansing was proven efficient. The timing of ingesting PEG-ELS is different between institutes and some ingest PEG-ELS as a whole at the night before colonoscopic examination and some ingested in split-dose manner which ingest half of the solution at previous night and remaining on the day of examination. Some institutes ask examinee to receive lavage solution on the day of examination. The manufacturer advices start taking medication on the day before the investigation according to their printed instruction on the package of PEG-ELS. Though there were a lot of studies that conducted to describe the result of colon cleansing in different fashion, the result is still controversial. This prospective, randomized, single-blinded trail evaluated and compared the efficacy of colon preparation at two timing of colon preparation, namely, in previous night or on the day of colonoscopic examination. In this study, we enrolled those who have already colon neoplasia detected during voluntary routine health check-up and received second colonoscopic examination for either elective polypectomy or endoscopic mucosectomy (EMR). We used not only the cleansing condition as a reference of adequate preparation; we also compared the diagnostic yield of lesion number as an objective comparator between these two methods.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the leading cause of cancer death not only in the Western countries but also in Taiwan. It is now the third leading cause of cancer mortality both in men and women in Taiwan. Previous studies revealed early detection of adenomatous polyp, the precursor lesion of CRC, plays a pivotal role in CRC prevention and removal of these lesions was proven to reduce CRC mortality. Fecal occult blood test (FOBT) is now the standard mass screening modality and colonoscopy is the standard procedure of choice if FOBT was positive. Nevertheless, colonoscopy is now gradually accepted as one of the powerful tool for colorectal cancer screening. Not only for survey after positive fecal test, it is also applied as primary screening modality for CRC screening.Colon cleansing before colonoscopy thus becomes critically important and inadequate preparation may lead to low diagnostic yield with missed lesions, increased risk of complication and prolonged procedure time. Though the importance of good colon preparation can not be over-emphasized, diet control before colonoscopy and ingestion of large amount of lavage solution remain a significant hurdle to overcome and investigators continue to seek for the ideal colon preparation with respect to quality and examinee satisfaction.

After the introduction of polyethylene glycol electrolyte lavage solution (PEG-ELS) for bowel preparation before colon procedures, its safety was well documented and the efficacy of colon cleansing was proven efficient. The timing of ingesting PEG-ELS is different between institutes and some ingest PEG-ELS as a whole at the night before colonoscopic examination and some ingested in split-dose manner which ingest half of the solution at previous night and remaining on the day of examination. Some institutes ask examinee to receive lavage solution on the day of examination. The manufacturer advices start taking medication on the day before the investigation according to their printed instruction on the package of PEG-ELS. Though there were a lot of studies that conducted to describe the result of colon cleansing in different fashion, the result is still controversial.

This prospective, randomized, single-blinded trail evaluated and compared the efficacy of colon preparation at two timing of colon preparation, namely, in previous night or on the day of colonoscopic examination. In this study, we enrolled those who have already colon neoplasia detected during voluntary routine health check-up and received second colonoscopic examination for either elective polypectomy or endoscopic mucosectomy (EMR). We used not only the cleansing condition as a reference of adequate preparation; we also compared the diagnostic yield of lesion number as an objective comparator between these two methods.

ELIGIBILITY:
Inclusion Criteria:

Those who had colon neoplasia detected at screening colonoscopy and requiring polypectomy or mucosectomy

Exclusion Criteria:

1. those who used anti-platelet agents or anticoagulants that can not be stopped,
2. those who had minute polyps detected that had been removed at screening colonoscopy,
3. those who had invasive cancer that require surgical intervention,
4. those who cannot complete total colonoscopy for any reason at health check-up.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Cleansing level of colon and detected lesion number during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Han-Mo Chiu, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan